## **CONSENT FORM**

Official Title: Evaluating the Effectiveness of the Occupational Therapy Handwriting Intervention Guideline on Handwriting Skills for Children: A Protocol for Clustered-Randomised Control Trial

Date of document: 1st October 2021



## **Consent Form**

Research project title: Evaluating the Effectiveness of the Occupational Therapy Handwriting Intervention Guideline on Handwriting Skills for Children

- I agree to participate in the research entitled Evaluating the Effectiveness of the Occupational Therapy Handwriting Intervention Guideline on Handwriting Skills for Children.
- I have read the information sheet related to the research study and understand the aims of the study.
- I am fully aware that I will remain anonymous throughout data reported and that I have the right to leave the study at any point.
- I am fully aware that data collected will be stored securely, safely and in accordance with Data Collection Act (1998).
- I am fully aware that I am not obliged to answer any question, but that I do so at my own free will.
- I agree to have my handwriting session to be recorded in video, so it can be evaluated for scoring purposes.

| SIGNATURE | <b>:</b> | | DATE : |
|------------|-------------|---|--------|
| NAME | : | | |
| RESEARCHER | R SIGNATURE | : | DATE : |

## For more information

This research has been reviewed and approved by the Research Ethics Board, Universiti Kebangsaan Malaysia. If you have any further questions or concerns about this study, please contact:

Mahfuzah binti Zainol Faculty of Health Sciences Universiti Kebangsaan Malaysia +6013-4740211 mahfuzah98@gmail.com You can also contact my supervisor: Dr. Masne binti Kadar

> Senior Lecturer Faculty of Health Sciences Universiti Kebangsaan Malaysia masne\_kadar@ukm.edu.my